CLINICAL TRIAL: NCT00983489
Title: Comparison of Impact of Breast Feeding Counseling of Mothers and Use of Audio-video Aids on Breast Feeding Rates at Six Weeks Postnatal Age
Brief Title: Comparison of Breast Feeding Counseling and Video Demonstration on Exclusive Breast Feeding Rates at 6 Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deen Dayal Upadhyay Hospital (Other)
Responsible Party: Principal Investigator, Dr Kanchan Sharma, DNB resident, Deen Dayal Upadhyay Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ddu001
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Results first posted 2013-05-24 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-04

CONDITIONS: Exclusive Breast Feeding
Keywords: breast feeding; counselling; video demonstration
MeSH Terms: conditions — Breast Feeding | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- counselling (Active Comparator): counselling: Breast feeding counselling will be done to mothers
  Interventions: Behavioral: counselling
- Video demonstration (Active Comparator): Video demonstration to mothers on the advantages of exclusive breast feeding
  Interventions: Behavioral: video demonstration
- Standard Care (No Intervention): Standard care includes the routine care provided to the neonates as per hospital protocol

INTERVENTIONS:
Behavioral: video demonstration — video will be shown to mothers
  Arms: Video demonstration
Behavioral: counselling — breast feeding counselling
  Arms: counselling

SUMMARY:
The investigators hypothesize that counseling of mothers will increase exclusive breast feeding rates at six weeks postnatal age. In developing countries like India,there is shortage of staff and the number of newborns cared is huge. So counseling of mothers for breast feeding becomes difficult. In such a situation using audio-visual aids may be a more practical option to increase breast feeding rates. Therefore the investigators will compare the use of video demonstration with counseling for exclusive breast feeding.

DETAILED DESCRIPTION:
1. Study design - Randomized controlled trial.
2. Inclusion criteria- All mothers who deliver at term at Deen Dayal Upadhayay Hospital [DDUH ]whether booked or unbooked.
3. Exclusion criteria -

   1. Sick mother who is unable to communicate
   2. Congenital malformation
   3. Babies admitted in neonatal intensive care unit
   4. HIV positive mother
   5. Mother on chemotherapy/planned for chemotherapy.
4. Setting of the study - The study will be conducted at postnatal wards of DDUH, New Delhi
5. Period of study-January 2009 to December 2009.
6. Sample size- We did a pilot study to see the baseline exclusive breast feeding rates at six weeks in mothers who delivered at DDUH. The baseline exclusive breast feeding rates at six weeks is 60%. Expecting a 10% absolute increase in exclusive breast feeding rates and alpha=0.05 and power beta=80% our sample size is 376 per group. Taking into account the loss to follow up of 20% we plan to enroll 470 mothers per group. So our sample size is 1410 mothers.
7. Ethics and consent-Ethical clearance will be obtained from ethical committee of DDUH. Written and informed consent will be taken from the mothers before enrolment.
8. Randomization - It will be an open-label randomized controlled trial. Random numbers will be obtained from a computer generated table. Mothers will be grouped into three groups: counseling group, video group and control group. The codes will be kept in sealed opaque envelopes. There will be allocation concealment since the mothers and the principle investigator will be unaware of the group to which they will be randomized.
9. Methods- The principle investigator will visit the postnatal wards daily except on holidays and look for the eligible mothers who will be asked for written and informed consent. Those who give the consent will be enrolled and randomized to counseling group, video group and control groups. The mothers in the intervention group will be counseled along with the husband and mother/mother-in-law/female caretaker. The mothers in the video group will be shown a video on breast feeding. The baseline characteristics of the three groups will be recorded. The mothers in the control group will receive standard care.

ELIGIBILITY:
Inclusion Criteria:

* All mothers who deliver at term at Deen Dayal Upadhayay Hospital [DDUH ]whether booked or unbooked.

Exclusion Criteria:

* Sick mother who is unable to communicate
* Congenital malformation
* HIV positive mother
* Mother on chemotherapy/planned for chemotherapy.

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1411 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2009 to June 2010 Tertiary care neonatal unit
Pre-assignment Details: None excluded after enrolment. Those who did not follow up were not analysed.
Period: Overall Study
Arm/Group | Counselling | Video Demonstration | Standard Care
Started | 511 | 453 | 447
Completed | 326 | 168 | 135
Not Completed | 185 | 285 | 312

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Counselling | Video Demonstration | Standard Care | Total
Number analyzed (Participants) | 511 | 453 | 447 | 1411
Age Continuous [Mean (Standard Deviation); unit: years] | 23.7 (3.2) | 23.9 (3.8) | 24.3 (3.6) | 24.0 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 243 | 215 | 219 | 677
  Male | 268 | 238 | 228 | 734
Region of Enrollment [Number; unit: participants]
  India | 511 | 453 | 447 | 1411

OUTCOME MEASURES:

1. Primary Outcome: Exclusive Breast Feeding Rate at Six Weeks Postnatal Age
Time Frame: 6 weeks
Measure: Number; unit: Participants
Arm/Group | Counselling | Video Demonstration | Standard Care
Number analyzed (Participants) | 326 | 168 | 135
Participants | 271 | 117 | 97

ADVERSE EVENTS:
Arm/Group | Counselling | Video Demonstration | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No